CLINICAL TRIAL: NCT00003546
Title: Phase II Chemoradiation Trial Using Gemcitabine in Patients With Locoregional Adenocarcinoma of the Pancreas
Brief Title: Gemcitabine Plus Radiation Therapy in Treating Patients With Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-89805; U10CA031946 (NIH); CLB-89805; CDR0000066601 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2004-09-13 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Pancreatic Cancer
Keywords: stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; adenocarcinoma of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Radiotherapy

ARMS (1):
- gemcitabine + radiation (Experimental): Patients receive radiation therapy 5 days per week for 5 1/2 weeks and gemcitabine IV over 30 minutes not greater than 2 hours prior to radiation therapy twice weekly. This combination radiation therapy and chemotherapy is followed by 2 weeks of rest. Patients with stable or responding disease receive a higher dose of gemcitabine IV over 30 minutes weekly for 3 weeks followed by 1 week of rest. This 4 week course is repeated 3 more times for a total of 16 weeks of gemcitabine therapy alone. Patients are followed every 2 months for the first year and then every 3 months for the next 2 years or until disease progression. Upon documentation of disease progression, patients are followed every 3 months for survival and secondary malignancy.
  Interventions: Drug: gemcitabine hydrochloride; Radiation: radiation therapy

INTERVENTIONS:
Drug: gemcitabine hydrochloride — given IV
Radiation: radiation therapy — 1.8 Gy to tumor bed

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy with radiation therapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of gemcitabine plus radiation therapy in treating patients with pancreatic cancer that cannot be removed surgically.

DETAILED DESCRIPTION:
OBJECTIVES: I. Estimate time to progression and overall survival of patients with locoregional adenocarcinoma of the pancreas treated with gemcitabine combined with radiation therapy. II. Estimate the biomarker response to this regimen through evaluation of circulating CA19-9 levels and correlate this response with survival of this patient population.

OUTLINE: Patients receive radiation therapy 5 days per week for 5 1/2 weeks and gemcitabine IV over 30 minutes not greater than 2 hours prior to radiation therapy twice weekly. This combination radiation therapy and chemotherapy is followed by 2 weeks of rest. Patients with stable or responding disease receive a higher dose of gemcitabine IV over 30 minutes weekly for 3 weeks followed by 1 week of rest. This 4 week course is repeated 3 more times for a total of 16 weeks of gemcitabine therapy alone. Patients are followed every 2 months for the first year and then every 3 months for the next 2 years or until disease progression. Upon documentation of disease progression, patients are followed every 3 months for survival and secondary malignancy.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study within 24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed adenocarcinoma of the pancreas Locoregional and not amenable to surgery based on 1 or more of the following: Size of pancreatic tumor greater than 5 cm Lymph nodes bulky, greater than 2 cm, but within radiation port Vascular involvement or impingement of major vessels (e.g., superior mesenteric artery, superior mesenteric vein, portal vein, hepatic artery) Involvement of colon (head lesions) or involvement of adrenal, kidney, or colon (tail lesions) Patients must be registered and begin treatment within 42 days of surgical staging No metastatic disease or nodal disease outside of radiation port documented by CT scan or MRI and chest x-ray

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Albumin greater than 3 g/dL Bilirubin less than 2.0 mg/dL Renal: Creatinine less than 2.0 mg/dL Calcium normal Other: No prior or concurrent malignancy within the past 5 years except inactive nonmelanoma skin cancer, carcinoma in situ of the cervix, or other curatively treated cancers Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior biologic therapy for carcinoma of the pancreas Chemotherapy: No prior chemotherapy for carcinoma of the pancreas No other concurrent chemotherapy Endocrine therapy: No prior endocrine therapy for carcinoma of the pancreas No concurrent hormone therapy (except for nondisease-related conditions) Radiotherapy: No prior radiation therapy for carcinoma of the pancreas No prior abdominal radiation therapy Surgery: See Disease Characteristics No prior surgery for carcinoma of the pancreas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 1998-09; Primary Completion 2003-12 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
progression free survival | up to 3 years
overall survival | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Margaret A. Tempero, MD, Study Chair — University of California, San Francisco
Locations (48):
- United States (48):
  - Veterans Affairs Medical Center - Birmingham, Birmingham, Alabama
  - University of California San Diego Cancer Center, La Jolla, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Vincent T. Lombardi Cancer Research Center, Georgetown University, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - University of Illinois at Chicago Health Sciences Center, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Veterans Affairs Medical Center - Togus, Togus, Maine
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Veterans Affairs Medical Center - Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Vermont Cancer Center, Burlington, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Result] Blackstock AW, Tepper JE, Niedwiecki D, Hollis DR, Mayer RJ, Tempero MA. Cancer and leukemia group B (CALGB) 89805: phase II chemoradiation trial using gemcitabine in patients with locoregional adenocarcinoma of the pancreas. Int J Gastrointest Cancer. 2003;34(2-3):107-16. doi: 10.1385/ijgc:34:2-3:107. PMID 15361643